CLINICAL TRIAL: NCT05039983
Title: Study of Epigallocatechin-3-gallate (EGCG) for Supportive and Symptomatic Management in Patients With Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, Principal Investigator, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTEEC2021
Record Dates: First submitted 2021-08-22; First posted 2021-09-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Obstruction
Keywords: EGCG; Esophageal obstruction; Supportive and Symptomatic Management
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EGCG application (Experimental): We have chosen a dose of 880 umol/L as the lower limit for this phase I study by referring to previous studies. Six dose levels for EGCG were defined as following: 880, 1760, 2640, 3430, and 4400 umol/L per dose. Dose escalation proceeded according to a standard phase I design with three patients initially treated on each tier. If, on any dose tier of EGCG, two of three patients or two of six patients experienced a more than grade II toxicity due to EGCG, dose escalation of EGCG would cease. The maximally tolerated dose (MTD) was defined as the highest dose with fewer than one-third of patients experiencing a dose-limiting toxicity (DLT) due to EGCG. EGCG solution was given continuously for 7 days before anti-tumor treatment.
  Interventions: Other: EGCG

INTERVENTIONS:
Other: EGCG — EGCG use various concentrations dissolved in 0.9% saline solution three times a day. A new batch is made up each time. For esophageal application, repeated swallowing of 30 ml of the EGCG solution is indispensable to assure the prolonged presence of drug the esophageal walls.

SUMMARY:
The main symptom of patients with advanced esophageal cancer is eating obstruction. In clinical practice, patients need to wait for a long time before anti-tumor treatment, which will lead to a rapid decline in the quality of life and nutritional status of patients, and severe patients sometimes need to place nasointestinal feeding tubes or endoscopic stents. EGCG has been shown to have antioxidant, anti-inflammatory and anti-tumor effects . The complex effects of EGCG may improve esophageal obstruction during the waiting period before antineoplastic therapy. The purpose of this phase I study was to explore the safety, recommended dose and preliminary efficacy of EGCG solution in the treatment of esophageal obstruction.

ELIGIBILITY:
Inclusion Criteria:

* confirmed pathological esophageal squamous cell carcinoma
* ≥18 years old
* the Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1
* no previous anti-tumor treatment
* no esophageal bleeding or fistula
* adequate hemocyte count, normal hepatic and renal functions
* Esophageal obstruction classified as grade 2 or grade 3 according to Stooler's dysphagia score

Exclusion Criteria:

* lactating or pregnant women
* known hypersensitivity or allergy to any kind green tea extract
* placement of small intestinal feeding tube or endoscopic stent treatment
* unable or refusing to take oral liquids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | baseline and up to 7 days post-treatment
  the toxicities will be reported by describing Adverse Events (AE) per CTCAE v5.0, by dose level, and type and grade of toxicity
Maximum tolerated dose (MTD) | baseline and up to 7 days post-treatment
  the toxicities will be reported by describing Adverse Events (AE) per CTCAE v5.0, by dose level, and type and grade of toxicity
Recommended phase 2 dose (RP2D) | baseline and up to 7 days post-treatment
  the toxicities will be reported by describing Adverse Events (AE) per CTCAE v5.0, by dose level, and type and grade of toxicity

SECONDARY OUTCOMES:
Imaging objective response rate | Change from Baseline esophageal stenosis size at 7 days
  Response rate of esophageal stenosis was determined by X-ray barium meal examination and/or contrast-enhanced CT
Symptom objective response rate | baseline and up to 7 days post-treatment
  choking and pain when swallowing was assessed by Stooler's dysphagia score and NRS
change in blood biochemical indicators | baseline and up to 8 days post-treatment
  This will be determined by prealbumin and albumin values

CONTACTS AND LOCATIONS:
Locations (1):
- Shan Dong cancer hospital and institute, Jinan, Shandong, China